CLINICAL TRIAL: NCT03625219
Title: Characterization of the Molecular Mechanisms Involved in Delayed-Type Hypersensitivity Reactions to House Dust Mite, Diphencyprone, Nickel, and Tuberculin Purified Protein Derivative in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovaderm Research Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Inno-6048
Record Dates: First submitted 2018-07-17; First posted 2018-08-10 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Delayed Type Hypersensitivity
MeSH Terms: conditions — Hypersensitivity, Delayed | interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: Cohort A Open label: 4 groups of 10 subjects Cohort B Double-Blind: 1 group of 20 subjects
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prednisone (Active Comparator): Cohort B only: Subjects will take 40 mg (8 x 5mg tablets) for three consecutive days, then 30 mg (6 x 5mg tablets), 20 mg (4 x 5 mg tablets), 10 mg (2 x 5 mg tablets) and 5 mg (1 x 5 mg tablet) daily for two consecutive days for each dose level for a total of 11 days of treatment.
  Interventions: Drug: Prednisone
- Placebo (Placebo Comparator): Cohort B only: 8 tablets for 3 consecutive days; then 6 tablets, 4 tablets, 2 tablets, and 1 tablet daily for 2 consecutive days for each tablet count for a total of 11 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisone — 40 mg (8 x 5mg tablets) for three consecutive days, then 30 mg (6 x 5mg tablets), 20 mg (4 x 5 mg tablets), 10 mg (2 x 5 mg tablets) and 5 mg (1 x 5 mg tablet) daily for two consecutive days for each dose level for a total of 11 days of treatment.
  Arms: Prednisone
Drug: Placebo — 8 tablets for 3 consecutive days; then 6 tablets, 4 tablets, 2 tablets, and 1 tablet daily for 2 consecutive days for each tablet count for a total of 11 days
  Arms: Placebo

SUMMARY:
This study will be conducted in 2 cohorts.

In Cohort A, approximately 40 subjects will participate in a single-center, open-label, non-randomized, parallel-group trial to investigate the molecular mechanisms involved in delayed-type hypersensitivity (DTH) to various antigens and assess the most appropriate skin challenge antigen to study the effect of systemic treatments on T cells.

Following evaluation of the results in Cohort A, approximately 20 healthy volunteers will be enrolled in Cohort B. This cohort will be a single-center, double-blind, randomized, two-arm, placebo-controlled study to evaluate the effect of corticosteroid treatment on the molecular and cellular phenotype of delayed hypersensitivity response to one if the antigens previously studied in Cohort A.

ELIGIBILITY:
Inclusion Criteria:

Cohort A:

* Subject is in good general health, according to the investigator's judgment based on vital signs, medical history, physical examination, and laboratory tests performed. For woman of childbearing potential, has had a negative urine pregnancy test at screening and on Day 1 (baseline).
* Subjects has acceptable reaction to selected antigens.
* Subject is willing to participate and is capable of giving informed consent. Note: Consent must be obtained prior to any study-related procedures.
* Subjects must be willing to comply with all study procedures and must be available for the duration of the study.

Cohort B:

* Subject is in good general health, according to the investigator's judgment based on vital signs, medical history, physical examination, and laboratory tests performed.
* For subject (woman) involved in any sexual intercourse that could lead to pregnancy, subject agrees that an effective contraceptive method will be used, from at least 4 weeks prior to screening until at least 4 weeks after the last study product administration. Effective contraceptive methods include hormonal contraceptives (combined oral contraceptive, patch, vaginal ring, injectable, or implant), intrauterine devices or intrauterine systems, vasectomized partner(s), tubal ligation, or a barrier method of contraception (male condom, female condom, cervical cap, diaphragm, contraceptive sponge) in conjunction with spermicide.

Note: Hormonal contraceptives must have been on a stable dose for at least 4 weeks before screening.

Note: The above list of contraceptive methods does not apply to subjects who are abstinent for at least 4 weeks before Day 1 and will continue to be abstinent from penile-vaginal intercourse throughout the study. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant.

Note: Women of nonchildbearing potential are defined as follows:

* Female who has had surgical sterilization (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy) or;
* Female who has had a cessation of menses for at least 12 months prior to screening without an alternative medical cause, and a follicle-stimulating hormone (FSH) test confirming nonchildbearing potential (refer to laboratory reference ranges for confirmatory levels).

  * For woman of childbearing potential, has had a negative urine and serum pregnancy test at screening and negative urine pregnancy test at Day 1 (baseline).
  * Subject is willing to participate and is capable of giving informed consent. Note: Consent must be obtained prior to any study-related procedures.
  * Subjects must be willing to comply with all study procedures and must be available for the duration of the study.

Exclusion Criteria:

Cohort A:

* Subject is a female who is breastfeeding, pregnant, or who is planning to become pregnant during the study.
* Subject has a known history of severe allergic reaction (local or systemic) to the tested hapten.
* Subject has a history of skin disease or presence of skin condition that, in the opinion of the investigator, would interfere with the study assessments including active urticaria, psoriasis, atopic dermatitis, active contact dermatitis and excited (angry back) skin syndrome.
* Medical history of dermatographism.
* History of contact dermatitis to medical adhesive bandages or glue.
* Presence of any scar tissue, tattoos, scratches, open sores, excessive hair, or skin damages at tested/injection sites that in the opinion of the investigator may interfere with study evaluations.
* Subject is known to have immune deficiency or is immunocompromised.
* Subject has a known history of chronic infectious disease (e.g., hepatitis B, hepatitis C, or infection with human immunodeficiency virus).
* Subject has evidence or suspicion of active or latent TB or a clear history of treatment for TB disease or infection
* Subject has a hypersensitivity to any of the components of the patch test matrix or the hapten excipients.
* Subject has a known hypersensitivity to Tuberculin Purified Protein Derivative or to any components of the formulation or container. .
* Subject previously had a severe reaction (e.g., necrosis, blistering, anaphylactic shock or ulcerations) to a previous tuberculin skin test

Cohort B:

* Subject is a female who is breastfeeding, pregnant, or who is planning to become pregnant during the study.
* Subject has a known history of severe allergic reaction (local or systemic) to the tested hapten.
* Subject has a history of skin disease or presence of skin condition that, in the opinion of the investigator, would interfere with the study assessments including active urticaria, psoriasis, atopic dermatitis, active contact dermatitis and excited (angry back) skin syndrome.
* Medical history of dermatographism.
* History of contact dermatitis to medical adhesive bandages or glue.
* Presence of any scar tissue, tattoos, scratches, open sores, excessive hair, or skin damages at tested/injection sites that in the opinion of the investigator may interfere with study evaluations.
* Subject is known to have immune deficiency or is immunocompromised.
* Subject has a known history of chronic infectious disease (e.g., hepatitis B, hepatitis C, or infection with human immunodeficiency virus).
* Subject has a contra-indication, or who would be at increased risk of adverse effects to systemic corticosteroid (e.g. active systemic fungal infection, extensive viral disease (such as measles, chickenpox and herpes simplex on the eye), diabetes, heart problems, peptic ulcer, inflammatory bowel disease, diverticulitis, active depression or psychosis, osteoporosis, cataracts, glaucoma, bleeding or clotting problems, high blood pressure, neurological problems, hypothyroidism, myasthenia, kidney diseases, liver diseases, history of low potassium or calcium in blood) that in the opinion of the investigator may put the subject at risk during the trial.
* Subject had a treated or non-treated systemic infection (bacterial or viral) within 4 weeks prior to screening until Day 1 (baseline).
* Subject has evidence or suspicion of active or latent TB or a clear history of treatment for TB disease or infection
* Subject received a live or live/attenuated vaccination within 4 weeks prior screening or intends to receive a live or live/attenuated vaccination during the course of the study.
* Subject has a positive result to the QuantiFERON-TB Gold test or Tuberculin Purified Protein Derivative (Mantoux) test (if applicable) at the screening visit.
* Subject has any clinically significant medical condition or physical/laboratory/ vital signs abnormality that would, in the opinion of the investigator, put the subject at undue risk or interfere with interpretation of study results.
* Use of any other concurrent medications known or suspected to interfere with study evaluations or that may pose a safety risk.
* Subject has a hypersensitivity to any of the components of the patch test matrix or the hapten excipients.
* Subject has a known hypersensitivity to Tuberculin Purified Protein Derivative or to any components of the formulation or container.
* Subject previously had a severe reaction (e.g., necrosis, blistering, anaphylactic shock or ulcerations) to a previous tuberculin skin test
* Subject has a known or suspected allergy or intolerance to excipients of the placebo.
* Subject has a known or suspected allergy to prednisone or any of its excipients or any other corticosteroids.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
Measurement of gene expression levels in skin biopsies following exposure to various antigens. | at least 4 days up to 18 days
  Measurement of gene expression levels in skin biopsies following exposure to various antigens.
Measurement of epidermal thickness in skin biopsies following exposure to various antigens. | at least 4 days up to 18 days
  Measurement of epidermal thickness in skin biopsies following exposure to various antigens.
Measurement of number of inflammatory cells in skin biopsies following exposure to various antigens. | at least 4 days up to 18 days
  Measurement of number of inflammatory cells in skin biopsies following exposure to various antigens.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, Principal Investigator — Principal Investigator
Locations (1):
- Innovaderm Research Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No